CLINICAL TRIAL: NCT03524092
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Arm, Placebo-Controlled Maintenance Study of Mirikizumab in Patients With Moderately to Severely Active Ulcerative Colitis (LUCENT 2)
Brief Title: A Maintenance Study of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: LUCENT 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16823; I6T-MC-AMBG (Other: Eli Lilly and Company); 2017-003238-96 (EudraCT Number)
Record Dates: First submitted 2018-05-10; First posted 2018-05-14 (Actual); Results first posted 2022-11-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
Keywords: Interleukin-23 (IL-23); IL-23p19; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Maintenance Period: Miri Induction Responder (IR) - Placebo (PBO) Subcutaneous (SC) (Placebo Comparator): Participants who were responders to blinded mirikizumab (miri) at Week 12 in induction study (LUCENT-1) randomized to withdraw from mirikizumab and start receiving PBO SC every 4 weeks (Q4W) from Week 0 of maintenance study (LUCENT-2) until Week 40 or until loss of response was confirmed.
  Interventions: Drug: Placebo SC
- Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC (Experimental): Participants who were responders to blinded mirikizumab at Week 12 in induction study (LUCENT-1) randomized to continue to receive 200 mg mirikizumab SC Q4W from Week 0 of LUCENT-2 until Week 40 or until loss of response was confirmed.
  Interventions: Drug: Mirikizumab SC
- Maintenance Period: PBO IR - PBO SC (Other): Participants who were responders to blinded placebo at Week 12 in induction study (LUCENT-1) continue to receive blinded placebo SC Q4W from Week 0 of LUCENT-2 until Week 40 or until loss of response was confirmed.
  Interventions: Drug: Placebo SC
- Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV (Other): Participants who received PBO SC or 200 mg mirikizumab SC Q4W during maintenance period and experienced a loss of response at or after Week 12, received rescue therapy with open label 300 mg mirikizumab intravenous (IV) Q4W for 3 doses.
  Interventions: Drug: Mirikizumab IV
- Extended Induction: Induction Nonresponders - 300mg Miri IV (Other): Participants who were nonresponders to blinded mirikizumab or placebo in induction study (LUCENT-1), received additional 3 doses of open label 300 mg mirikizumab IV Q4W during extended induction period from Week 0 of LUCENT-2 until Week 12.
  Interventions: Drug: Mirikizumab IV
- Open Label Maintenance: Delayed Responders - 200 mg Miri SC (Other): Participants who initially did not respond to induction study (LUCENT-1), but responded to extended induction therapy at Week 12 of LUCENT-2 (delayed responders), received 200 mg mirikizumab SC Q4W during open label maintenance period from Week 12 until Week 40.
  Interventions: Drug: Mirikizumab SC

INTERVENTIONS:
Drug: Mirikizumab SC — Administered SC
  Other Names: LY3074828
  Arms: Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC; Open Label Maintenance: Delayed Responders - 200 mg Miri SC
Drug: Mirikizumab IV — Administered IV
  Other Names: LY3074828
  Arms: Extended Induction: Induction Nonresponders - 300mg Miri IV; Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV
Drug: Placebo SC — Administered SC
  Arms: Maintenance Period: Miri Induction Responder (IR) - Placebo (PBO) Subcutaneous (SC); Maintenance Period: PBO IR - PBO SC

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mirikizumab as maintenance therapy in participants who completed as clinical responders in the prior 12-week induction study LUCENT-1 (NCT03518086).

ELIGIBILITY:
Inclusion Criteria:

* Have completed Study AMAN (NCT03518086), with at least 1 study drug administration and without early termination of study drug.
* Are willing and able to complete the scheduled study assessments, including endoscopy and daily diary entry.
* If female, must meet the contraception requirements.

Exclusion Criteria:

* Participants diagnosed with Crohn's disease or inflammatory bowel disease-unclassified (indeterminate colitis) during the induction study AMAN (NCT03518086).
* Participants with a bowel resection or other surgery for the treatment of UC during the previous induction study AMAN (NCT03518086), or are likely to require surgery for the treatment of UC during study AMBG.
* Participants with evidence of colonic dysplasia or have been diagnosed with cancer of the gastrointestinal tract during study AMAN (NCT03518086).
* Participants diagnosed with clinically important infection including, but not limited to, hepatitis B, hepatitis C, HIV/AIDS, and active tuberculosis (TB) during the induction study AMAN (NCT03518086).
* Participants who initiate a new prohibited medication during the induction study AMAN (NCT03518086).
* Participants with certain laboratory abnormalities prior to start of AMBG that would require permanent discontinuation from study drug.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2025-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (384):
- United States (57):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Dcr-Pi, Pc, Litchfield Park, Arizona
  - Maricopa Integrated Health System, Phoenix, Arizona
  - Physicians Research Group, Tempe, Arizona
  - Valley Gastroenterology, Arcadia, California
  - Care Access Research, Berkeley, California
  - Om Research, LLC, Lancaster, California
  - California Medical Research Associates, Northridge, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - Direct Helpers Research Center, Hialeah, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - SIH Research, LLC, Kissimmee, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Center for Interventional Endoscopy, Orlando, Florida
  - Clintheory Healthcare, Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Florida Medical Clinic LLC, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - NorthShore University HealthSystem, Evanston, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Delta Research Partners LLC, Monroe, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - MNGI Digestive Health - Plymouth Endoscopy Center & Clinic, Plymouth, Minnesota
  - Care Access Research LLC, Jackson, Mississippi
  - Digestive Health Specialists, Tupelo, Mississippi
  - Northwell Health, Great Neck, New York
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina Center for Inflammatory Bowel Disease, Chapel Hill, North Carolina
  - Carolina Digestive Diseases and Endoscopy Center, Greenville, North Carolina
  - Paramount Medical Research, Middleburg Heights, Ohio
  - Care Access - Youngstown, Poland, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Digestive Disease Associates, Wyomissing, Pennsylvania
  - Midwest Medical Care, Sioux Falls, South Dakota
  - Gastro One, Germantown, Tennessee
  - Galen Medical Group, Hixson, Tennessee
  - Digestive Health Associates of Texas, Garland, Texas
  - Houston Methodist Research Ins, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Care Access Research LLC - Salt Lake City, Ogden, Utah
  - Emeritas Research Group, Leesburg, Virginia
  - The Gastroenterology Group, P.C., Reston, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Argentina (7):
  - Centro de Investigaciones Metabólicas (CINME), CABA, Buenos Aires
  - Mautalen Salud e Investigacion-Centro de Osteopatías Médicas, Ciudad Autonoma de Buenos Air, Buenos Aires
  - CER Instituto Medico, Quilmes, Buenos Aires
  - Fundación de Estudios Clínicos, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - C.I.C.E. 9 de Julio, San Miguel de Tucumán, Tucumán Province
  - Hospital Privado Centro Medico de Cordoba SA, Córdoba
- Australia (8):
  - Princess Alexandra Hospital, Harlow, Essex
  - Coastal Digestive Health, Maroochydore, Queensland
  - Mater University Hospital, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital Outpatients, Box Hill, Victoria
  - Melbourne Gastrointestinal Investigation Unit (MGIU), Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Austria (3):
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitätsklinikum Salzburg, Salzburg
  - Medical University of Vienna, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - Centre Hospitalier de Wallonie Picarde - Site Notre Dame, Tournai, Wallonne, Région
  - AZ Klina, Brasschaat
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (9):
  - West Edmonton Diabetes Center, Edmonton, Alberta
  - The Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - PerCuro Clinical Research, Victoria, British Columbia
  - Victoria Hospital, London, Ontario
  - University of Western Ontario, London, Ontario
  - Centre de santé et de services sociaux Champlain-Charles-Le Moyne, Greenfield Park, Quebec
  - Hopital Maisonneure-Rosemount, Montreal, Quebec
  - Inflammatory Bowel Disease Centre Montreal General Hospital - MUHC, Montreal, Quebec
- China (28):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Xiangya Hospital Central South University, Kaifu District, Changsha City
  - The Affiliated 2nd Hosp. of Third Military Med. Univ. of PLA, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nanjing Medical University - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Jilin Central General Hospital, Jilin, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Taian City Central Hospital, Taian, Shandong
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Renji Hospital Affliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Kunming Medical College Affiliated First Hospital, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second Affiliated Hospital of Zhejiang University School of Med, Hangzhou, Zhejiang
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital YuYing Childens Hospital of Wenzhou Medical university, Wenzhou, Zhejiang
  - Tongji Hospital of Tongji University, Wuhan
- Czechia (9):
  - Vojenská Nemocnice Brno, Brno, Brno-město
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Hl. M. Praha
  - Hepato-Gastroenterologie HK, Hradec Králové, Hradec Králové
  - MUDr. Gregar, s.r.o., Olomouc, Olomoucký kraj
  - A-Shine, Pilsen, Plzeň-město
  - MEDIENDO, Prague, Praha 8
  - Fakultni Nemocnice u sv. Anny v Brne, Brno
  - PreventaMed, s.r.o., Olomouc
  - ISCARE Clinical Centre, Prague
- Denmark (2):
  - Herlev and Gentofte Hospital, Herlev
  - Zealand University Hospital Køge, Køge
- France (15):
  - Hopital de Hautepierre - Service d'Hépatogastroentérolgie, Strasbourg, Bas Rhin
  - Hopital Saint-Louis, Paris, Cedex 10
  - CHU Lille - Hôpital Claude Huriez, Lille, Nord
  - Hôpital Beaujon, Clichy, Paris
  - Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -, Pierre-Bénite, Rhone
  - CHU Amiens Picardie-Site Sud - RDC Service Hépato gastro, Amiens, Somme
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - CHRU de Montpellier-Hopital St Eloi, Montpellier
  - Hopital L'Archet 2, Nice
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Robert Debre Hospital, Reims
  - CHU de Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - CHRU Nancy Brabois - Hôpital d'Enfants, Vandœuvre-lès-Nancy
- Germany (9):
  - Medizinische Hochschule Hanover, Hanover, Lower Saxony
  - Gemeinschaftspraxis Dr. Peter Uebel, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle, Saxony-Anhalt
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Charité Campus Virchow-Klinikum, Berlin
  - Krankenhaus Waldfriede, Berlin
  - Städtisches Klinikum Brandenburg, Brandenburg
  - HaFCED - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - Internistische Praxisgemeinschaft, Weyhe
- Hungary (9):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred, EU
  - Jávorszky Ödön Kórház, Vác, Pest County
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis Egyetem, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Endomedix Diagnosztikai Központ - Miskolc, Miskolc
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont I. Belgyogyaszati Klinika, Szeged
  - CLINFAN Szolgáltató Kft, Szekszárd
- India (14):
  - Centre for Liver Research & Diagnostics, Deccan College of Medical Sciences, Owaisi Hospital & Research Centre, Hyderabad, Andhra Pradesh
  - Apollo Research and Innovations, Apollo Hospitals International Ltd, Gandhinagar, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujarat
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Bangalore Medical College and Research Institute, Bangalore, Karnataka
  - M S Ramaiah Medical College and Hospitals, Bangalore, Karnataka
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur, Maharashtra
  - Poona Medical Foundation. Ruby Hall Clinic, Pune, Maharashtra
  - Datta Meghe Institute of Medical Sciences (DU), Acharya Vinoba Bhave Rural Hospital, Wardha, Maharashtra
  - Escorts Heart Institute and Research Centre Ltd, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Gandhi Hospital, Hyderabad, Telangana
  - King George Medical University, Lucknow, Uttar Pradesh
- Beaumont Hospital, Dublin, Dublin, Ireland
- Israel (6):
  - Shaare Zedek Medical Center, Bait Vagan, Jerusalem
  - Soroka Medical Center - Pediatric Outpatient Clinic, Beersheba
  - Galilee Medical Center Department of Internal Medicine A, Nahariya
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - King Fahad Medical City, Ẕerifin
- Italy (14):
  - Presidio di Rho, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Istituti di Ricovero e Cura a Carattere Scientifico Policlinico San Donato Gastroenterologia, San Donato Milanese, Milano
  - Ospedale Sandro Pertini, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Torre, Roma
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda ospedaliero-universitaria Mater Domini, Catanzaro
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Gastroenterology and Endoscopy Unit IRCCS Ca' Granda Ospedale Maggiore Policlinico Foundation, Milan
  - Azienda Ospedaliera Universitaria Policlinico de Modena, Modena
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Policlinico Gemelli - Università Cattolica del Sacro Cuore, Roma
  - Ospedale Mauriziano Umberto I, Torino
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia Gastroenterologia, Udine
- Japan (48):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi, Fukoka
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Hidaka Coloproctology Clinic, Kurume-shi, Fukuoka
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Takasaki General Medical Centar, Takasaki, Gunma
  - NHO Mito Medical Center, Ibaraki-machi, HigaShiibaraki-Gun
  - Asahikawa City Hospital, Asahikawa, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Aoyama Clinic GI Endoscopy & IBD Center, Kobe, Hyōgo
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Ofuna Central Hospital, Kamakura, Kanagawa
  - Kawasaki Municipal Hospital, Kawasaki, Kanagawa
  - Sankikai Yokohama Shin midori General Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Showa University Northern Yokohama Hospital, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Mie University Hospital, Tsu, Mie-ken
  - Takagi Clinic - Sendai, Sendai, Miyagi
  - Nagaoka Chuo General Hospital, Nagaoka-shi, Niigata
  - Ishida Clinic of IBD and Gastroenterology, Ōita, Oita Prefecture
  - Sai Gastroenterologist Proctology, Fujiidera, Osaka
  - Infusion Clinic, Osaka, Osaka
  - NHO Osaka National Hospital, Osaka, Osaka
  - Saga-Ken Medical Center Koseikan, Saga, Saga-ken
  - Kumagaya General Hospital, Kumagaya-shi, Saitama
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyō, Tokyo
  - Showa University Koto Toyosu Hospital, Koto-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-Ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - JHCO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo-To
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-ku, Tokyo-To
  - Fukuoka University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Sameshima Hospital, Kagoshima
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Okayama University Hospital, Okayama
  - Tokitokai Tokito Clinic, Saitama
  - Toyama Prefectural Central Hospital, Toyama
- Latvia (3):
  - Pauls Stradins Clinical Univeristy Hospital, Riga, Rīga
  - Digestive Diseases Center "Gastro", Riga
  - Riga Eastern Clinical University Hospital, Riga
- Lithuania (5):
  - Respublikine Panevezio ligonine, Panevezys, Panevėžys
  - Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas
  - Republic Hospital of Klaipeda, Klaipėda
  - Klaipeda Seamen's Hospital, Klaipėda
  - Vilnius University Hospital Santariskiu Clinics, Vilnius
- Malaysia (3):
  - Universiti Sains Malaysia, Kubang Kerian, Kelantan
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Ampang, Ampang, Selangor
- Mexico (5):
  - Investigación Biomédica para el Desarrollo de Fármacos S.A. de C.V., Zapopan, Jalisco
  - Centro de Investigación Clínica Acelerada, Mexico City, Mexico City
  - Centro Para el Desarrollo de la Medicina y de Asistencia Medica S.C, Culiacán, Sinaloa
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Sociedad de Metabolismo y Corazon, Veracruz
- Netherlands (4):
  - St Elisabeth Ziekenhuis, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC, Amsterdam, North Holland
  - Bernhoven Ziekenhuis, Uden
  - UMC Utrecht, Dept. of Internal Medicine, MDL, Utrecht
- Poland (20):
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Topolowa Medicenter, Krakow, Lesser Poland Voivodeship
  - Medicenter Nowy Targ, Nowy Targ, Lesser Poland Voivodeship
  - NZOZ Formed, Wadowice, Lesser Poland Voivodeship
  - LexMedica, Wroclaw, Lower Silesian Voivodeship
  - ZOZ Gastromed, Lublin, Lublin Voivodeship
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - NZOZ Vivamed, Warsaw, Masovian Voivodeship
  - Promedica Dental Clinic, Będzin, Silesian Voivodeship
  - SONOMED Centrum Medyczne, Szczecin, West Pomeranian Voivodeship
  - All-Medicus, Katowice
  - Wojewodzki Specjalistyczny Szpital w Olsztynie, Olsztyn
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - Gastromed Kopoń Zmudziński I Wspólnicy Spółka Jawna Specjalistyczne Centrum Gastrologii I Endoskopii, Torun
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Zdrowia MDM, Warsaw
  - Centrum Medyczne NeuroProtect, Warsaw
  - PlanetMed Sp.z o.o., Wroclaw
  - ETG Zamość, Zamość
  - KO-Med Centrum Medyczne, Straszów, Świętokrzyskie Voivodeship
- Romania (6):
  - CCBR Clinical Research, Bucharest, București
  - MedLife Grivita, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Hifu Terramed Conformal SRL, Bucharest
  - Spital Pelican Oradea, Oradea
- Russia (25):
  - Scientific Centre of Reconstructive and Restorative Surgery, Irkutsk, Irkutsk Oblast
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk, Kareliya, Respublika
  - Nizhny Novgorod Regional Hospital N.A. Semashko, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Private Healthcare Institution Clinical Hospital Russian Railways - Medicine of Nizhniy Novgorod, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Novosibirski Gastrocenter, Novosibirsk, Novosibirsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - Scientific research center ECO-security, Saint Petersburg, Sankt-Peterburg
  - Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - Medical and Sanitary Division of Severstal, Cherepovets
  - Alliance Biomedical URAL Group, Izhevsk
  - Clinical Trials Center of Medical Institute, Kaliningrad
  - State Autonomous Institution of Healthcare "Republican Clinical Hospital of the Ministry of Healthcare of Republic Tatarstan, Kazan'
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo
  - Medical rehabilitation center, Moscow
  - LLC "Medicine Center SibNovoMed", Novosibirsk
  - Clinical Diagnostic Center Ultramed, Omsk
  - City Mariinskaya Hospital, Saint Petersburg
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Non-state Healthcare Institution "Roadway Clinical Hospital of OJSC Russian Railways, Saint Petersburg
  - Saint Petersburg State Medical University n.a. Pavlov I.P., Saint Petersburg
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - Medical Institute REAVIZ, Samara
  - Stavropol State Medical University, Stavropol
  - Yaroslavl Municipal HI Clinical Hospital #8, Yaroslavl
  - LLC MA New Hospital, Yekaterinburg
- Serbia (6):
  - Clinical Hospital Center Zvezdara, Belgrade, Beograd
  - University Medical Center "Bezanijska kosa", Belgrade, NAP
  - Regional Hospital Dr Radivoj Simonovic Sombor, Sombor, Vojvodina
  - Sremska Mitrovica Health Centre, Sremska Mitrovica, Vojvodina
  - General Hospital "Djordje Joanovic", Zrenjanin, Vojvodina
  - Clinical Center Kragujevac Gastroenterohepatology Clinic, Kragujevac
- Slovakia (5):
  - KM Management, Nitra, Nitra Region
  - Gastro, Prešov, Presov
  - Endomed, s.r.o., Vranov N. Toplou, Presov
  - Fakultna nemocnica s poliklinikou Roosevelta Banska Bystrica, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Bratislava
- South Korea (9):
  - Severance Hospital, Yonsei University Health System, Wŏnju, Gangwon-do
  - Kyung Hee University Hospital, Seoul, Korea
  - Dong-A University Hospital, Busan, Pusan-Kwangyǒkshi
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon, Taejǒn-Kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Busan
  - Yeungnam Univeristy Medical Center, Daegu
- Spain (12):
  - Hospital Universitario Virgen Del Rocio, Seville, Andalusia
  - Hospital Universitari Son Espases, Palma de Mallorca, Baleares Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital De Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Gen. Juan Ramon Jimenez - Depto de Digestivo, Sagunto, Valencia
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Instituto de Ciencias Médicas, Alicante
  - Hospital Universitari de Girona, Girona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
- Switzerland (4):
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern, Canton of Bern
  - Inselspital Bern, Bern
  - Kantonsspital St.Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - Health management center, Taipei
- Turkey (Türkiye) (5):
  - Antalya Egitim ve Arastırma Hastanesi, Kocaeli, Antalya
  - Acibadem Universitesi - Acibadem Kozyatagi Hastanesi, Kadıköy, Istanbul
  - Kocaeli University Medical Faculty Hospital, İzmit, Kocaeli
  - Mersin University Medical Faculty, Yenişehir, Mersin
  - Ege Universitesi Hastanesi, Izmir
- Ukraine (21):
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - City Clinical Hospital No. 2, Kharkiv, Kharkivs’ka Oblast’
  - Kherson City Clinical Hospital, Kherson, Kherson Oblast
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev, Kyiv Oblast
  - Lviv Railway Clinical Hospital, Lviv, Lviv Oblast
  - Lviv Regional Endocrinology Dispensary, Lviv, Lviv Oblast
  - Municipal non-profit enterprise "Lviv Territorial Medical Union "Multidisciplinary Clinical Hospital of Em -T, Lviv, Lviv Oblast
  - Poltova Oblast Clinical Hospital IM.M.V.Sklifosovskoho, Poltava, Poltava Oblast
  - Diaservis - Medical and Diagnostic Center, Zaporizhia, Zaporizhzhia Oblast
  - Kharkiv City Student Hospital, Kharkiv
  - GI L.T. Malaya TI Namsu, Kharkiv
  - Treatment-Diagnostic Center of Private Enterprise of PPC Atsynus, Kropyvnytskyi
  - Kyiv Municipal Clinical Hospital #1, Kyiv
  - Communal institution of the Kyiv Regional Council "Kyiv Regional Clinical Oncology Dispensary", Kyiv
  - Communal Enterprise "Odesa Regional Clinical Hospital", Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Vinnytsia RCH of Veterans of War Dept of Therapy#1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - M.I. Pyrogov Regional Clinical Hospital, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Communal Institution of Kyiv Regional Council Kyiv Regional Hospital #2, Zaporizhzhia
- United Kingdom (6):
  - Queens Hospital, Romford, Essex
  - Fairfield General Hospital, Bury, Great Britain
  - St Thomas' Hospital, Great Maze Pond, London
  - Whipps Cross University Hospital, London, Surrey
  - Morriston Hospital, Swansea, Swansea [Abertawe Gb-ata]
  - St James's University Hospital, Leeds, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Clemow DB, Dubinsky MC, Baygani SK, Sands BE, Keohane A, Danese S, Schreiber S, Walsh AJ, Hibi T, Gibble TH, Moses RE, Travis SPL. Bowel urgency in ulcerative colitis: effect of baseline urgency and change in urgency in response to mirikizumab. J Patient Rep Outcomes. 2025 Jul 1;9(1):75. doi: 10.1186/s41687-025-00906-0. PMID 40591171
- [Derived] Panaccione R, Chan-Diehl F, Baygani S, Fisher DA, Moses RE, Siegmund B, Walsh A, Kobayashi T, Dulai PS, Travis S. Fecal Calprotectin and C-Reactive Protein Association With Histologic and Endoscopic Endpoints in Mirikizumab-Treated Patients With Ulcerative Colitis. Crohns Colitis 360. 2025 Jun 14;7(2):otaf043. doi: 10.1093/crocol/otaf043. eCollection 2025 Apr. PMID 40589947
- [Derived] Lee SD, Ehrlich AC, Pellanda P, Kaiser C, Todd K, Moses R, Walsh A. Long-Term Safety of Mirikizumab in Patients With Moderately to Severely Active Ulcerative Colitis: An Integrated 2-Year Safety Analysis. Am J Gastroenterol. 2025 Dec 1;120(12):2857-2866. doi: 10.14309/ajg.0000000000003407. Epub 2025 Mar 12. PMID 40071779
- [Derived] Sands BE, D'Haens G, Clemow DB, Irving PM, Johns JT, Gibble TH, Abreu MT, Lee SD, Hisamatsu T, Kobayashi T, Dubinsky MC, Vermeire S, Siegel CA, Peyrin-Biroulet L, Moses RE, Milata J, Panaccione R, Dignass A. Three-Year Efficacy and Safety of Mirikizumab Following 152 Weeks of Continuous Treatment for Ulcerative Colitis: Results From the LUCENT-3 Open-Label Extension Study. Inflamm Bowel Dis. 2025 Jul 7;31(7):1876-1890. doi: 10.1093/ibd/izae253. PMID 39448057
- [Derived] Danese S, Dignass A, Matsuoka K, Ferrante M, Long M, Redondo I, Moses R, Maier S, Hunter Gibble T, Morris N, Milch C, Abreu MT. Early and Sustained Symptom Control with Mirikizumab in Patients with Ulcerative Colitis in the Phase 3 LUCENT Programme. J Crohns Colitis. 2024 Nov 4;18(11):1845-1856. doi: 10.1093/ecco-jcc/jjae088. PMID 38869019
- [Derived] Long MD, Schreiber S, Hibi T, Gibble TH, Fisher DA, Park G, Moses RE, Higgins PDR, Lindsay JO, Lee SD, Escobar R, Jairath V. Association of Bowel Urgency With Quality-of-Life Measures in Patients With Moderately-to-Severely Active Ulcerative Colitis: Results From Phase 3 LUCENT-1 (Induction) and LUCENT-2 (Maintenance) Studies. Crohns Colitis 360. 2024 Jan 6;6(1):otae001. doi: 10.1093/crocol/otae001. eCollection 2024 Jan. PMID 38313767
- [Derived] Sands BE, Feagan BG, Hunter Gibble T, Traxler KA, Morris N, Eastman WJ, Schreiber S, Jairath V, Long MD, Armuzzi A. Mirikizumab Improves Quality of Life in Patients With Moderately-to-Severely Active Ulcerative Colitis: Results From the Phase 3 LUCENT-1 Induction and LUCENT-2 Maintenance Studies. Crohns Colitis 360. 2023 Nov 7;5(4):otad070. doi: 10.1093/crocol/otad070. eCollection 2023 Oct. PMID 38034882
- [Derived] Chua L, Friedrich S, Zhang XC. Mirikizumab Pharmacokinetics in Patients with Moderately to Severely Active Ulcerative Colitis: Results from Phase III LUCENT Studies. Clin Pharmacokinet. 2023 Oct;62(10):1479-1491. doi: 10.1007/s40262-023-01281-z. Epub 2023 Aug 23. PMID 37610533
- [Derived] D'Haens G, Dubinsky M, Kobayashi T, Irving PM, Howaldt S, Pokrotnieks J, Krueger K, Laskowski J, Li X, Lissoos T, Milata J, Morris N, Arora V, Milch C, Sandborn W, Sands BE; LUCENT Study Group. Mirikizumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2023 Jun 29;388(26):2444-2455. doi: 10.1056/NEJMoa2207940. PMID 37379135
- [Derived] Magro F, Pai RK, Kobayashi T, Jairath V, Rieder F, Redondo I, Lissoos T, Morris N, Shan M, Park M, Peyrin-Biroulet L. Resolving Histological Inflammation in Ulcerative Colitis With Mirikizumab in the LUCENT Induction and Maintenance Trial Programmes. J Crohns Colitis. 2023 Oct 20;17(9):1457-1470. doi: 10.1093/ecco-jcc/jjad050. PMID 37057827
- See also: A Maintenance Study of Mirikizumab in Participants With Moderately to Severely Active Ulcerative Colitis (LUCENT 2) — https://trials.lillytrialguide.com/en-US/trial/6R2qUhQWcgImGasYaaGmYq

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1177 Participants enrolled in the study of which 716 participants entered to Blinded Maintenance Period as Induction Responder (IR) and 461 participants entered into open label extended Induction period as Induction Nonresponders.
Pre-assignment Details: This study was designed to evaluate the safety and efficacy of mirikizumab (miri) in achieving remission at Week (Wk) 40 in participants who completed the 12-week induction study I6T-MC-AMAN (NCT03518086) as clinical responders to mirikizumab. Results for maximum extended enrollment (ME2) participants will be posted after the study completion.
Groups:
- Maintenance Period: Miri IR - Placebo (PBO) Subcutaneous (SC): Participants who were responders to blinded mirikizumab (miri) at Week 12 in induction study (LUCENT-1) randomized to withdraw from mirikizumab and start receiving PBO SC every 4 weeks (Q4W) from Week 0 of maintenance study (LUCENT-2) until Week 40 or until loss of response was confirmed.
- Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV: Participants who received blinded PBO SC or blinded 200 mg mirikizumab SC Q4W during maintenance period and experienced a loss of response at or after Week 12, received rescue therapy with open label 300 mg mirikizumab intravenous (IV) Q4W for 3 doses.
- Open Label Maintenance: Delayed Responders - 200 mg Miri SC: Participants who initially did not respond to induction study (LUCENT-1), but responded to extended induction therapy at Week 12 of LUCENT-2 (delayed responders), received 200 mg mirikizumab SC Q4W during open label maintenance period from Week 12 until Week 40 or until early termination (rescue was not available for these participants).
Period: Blinded Maintenance Period (Wk 0-40)
Arm/Group | Maintenance Period: Miri IR - Placebo (PBO) Subcutaneous (SC) | Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC | Maintenance Period: PBO IR - PBO SC | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV | Extended Induction: Induction Nonresponders - 300mg Miri IV | Open Label Maintenance: Delayed Responders - 200 mg Miri SC
Started | 192 | 389 | 135 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 192 | 389 | 135 | 0 | 0 | 0
Completed | 119 | 347 | 90 | 0 | 0 | 0
Not Completed | 73 | 42 | 45 | 0 | 0 | 0
Not completed — Adverse Event | 16 | 6 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 8 | 6 | 7 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 8 | 6 | 0 | 0 | 0
Not completed — Loss of Response Rescue Period | 42 | 19 | 29 | 0 | 0 | 0
Period: Loss of Response Rescue Period
Arm/Group | Maintenance Period: Miri IR - Placebo (PBO) Subcutaneous (SC) | Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC | Maintenance Period: PBO IR - PBO SC | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV | Extended Induction: Induction Nonresponders - 300mg Miri IV | Open Label Maintenance: Delayed Responders - 200 mg Miri SC
Started | 0 (Participants were assigned to this arm only after at least 12 weeks of blinded maintenance period.) | 0 (Participants were assigned to this arm only after at least 12 weeks of blinded maintenance period.) | 0 (Participants were assigned to this arm only after at least 12 weeks of blinded maintenance period.) | 90 (Included only participants who experienced loss of response and were eligible for loss of response rescue induction.) | 0 | 0
Completed | 0 | 0 | 0 | 81 | 0 | 0
Not Completed | 0 | 0 | 0 | 9 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 5 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Period: Open Label Extended Induction (Wk 0-12)
Arm/Group | Maintenance Period: Miri IR - Placebo (PBO) Subcutaneous (SC) | Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC | Maintenance Period: PBO IR - PBO SC | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV | Extended Induction: Induction Nonresponders - 300mg Miri IV | Open Label Maintenance: Delayed Responders - 200 mg Miri SC
Started | 0 | 0 | 0 | 0 (Participants were assigned to this arm only during loss of response rescue period.) | 461 (Included only participants who entered open label extended induction period.) | 0
Completed | 0 | 0 | 0 | 0 | 271 | 0
Not Completed | 0 | 0 | 0 | 0 | 190 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 11 | 0
Not completed — Covid-19 related study disruption | 0 | 0 | 0 | 0 | 4 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 162 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 6 | 0
Not completed — Lack of capacity due to lack of staff | 0 | 0 | 0 | 0 | 1 | 0
Period: Open Label Maintenance Period (Wk 12-40)
Arm/Group | Maintenance Period: Miri IR - Placebo (PBO) Subcutaneous (SC) | Maintenance Period: Miri IR - 200 Milligram (mg) Miri SC | Maintenance Period: PBO IR - PBO SC | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV | Extended Induction: Induction Nonresponders - 300mg Miri IV | Open Label Maintenance: Delayed Responders - 200 mg Miri SC
Started | 0 | 0 | 0 | 0 | 0 (Participants were assigned to this arm only during open label extended induction period.) | 271 (Included only participants who entered open label maintenance period.)
Completed | 0 | 0 | 0 | 0 | 0 | 256
Not Completed | 0 | 0 | 0 | 0 | 0 | 15
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Covid-19 related study disruption | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Maintenance Period: Miri IR - PBO SC: Participants who were responders to blinded mirikizumab (miri) at Week 12 in induction study (LUCENT-1) randomized to withdraw from mirikizumab and start receiving PBO SC every 4 weeks (Q4W) from Week 0 of maintenance study (LUCENT-2) until Week 40 or until loss of response was confirmed.
- Maintenance Period: Miri IR - 200 mg Miri SC: Participants who were responders to blinded mirikizumab at Week 12 in induction study (LUCENT-1) randomized to continue to receive 200 mg mirikizumab SC Q4W from Week 0 of LUCENT-2 until Week 40 or until loss of response was confirmed.
- Total: Total of all reporting groups
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC | Maintenance Period: PBO IR - PBO SC | Extended Induction: Induction Nonresponders - 300mg Miri IV | Total
Number analyzed (Participants) | 192 | 389 | 135 | 461 | 1177
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.20 (12.88) | 43.30 (14.13) | 40.80 (13.40) | 43.40 (13.86) | 42.70 (13.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 160 | 61 | 166 | 465
  Male | 114 | 229 | 74 | 295 | 712
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data collected only for United States (US) participants.
  Participants
    Hispanic or Latino | 2 | 12 | 2 | 11 | 27
    Not Hispanic or Latino | 18 | 33 | 8 | 53 | 112
    Unknown or Not Reported | 172 | 344 | 125 | 397 | 1038
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 2 | 4 | 10
  Asian | 51 | 93 | 28 | 87 | 259
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 6 | 0 | 6 | 12
  White | 138 | 285 | 103 | 358 | 884
  More than one race | 0 | 0 | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 0 | 4 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 5 | 0 | 5 | 11
  Australia | 0 | 3 | 0 | 9 | 12
  Austria | 2 | 2 | 0 | 4 | 8
  Belgium | 1 | 2 | 2 | 4 | 9
  Canada | 3 | 5 | 2 | 21 | 31
  China | 3 | 4 | 1 | 7 | 15
  Czechia | 7 | 19 | 11 | 15 | 52
  Denmark | 3 | 3 | 0 | 1 | 7
  France | 10 | 18 | 6 | 23 | 57
  Germany | 5 | 13 | 3 | 16 | 37
  Hungary | 1 | 8 | 2 | 12 | 23
  India | 18 | 25 | 16 | 13 | 72
  Ireland | 0 | 1 | 0 | 0 | 1
  Israel | 3 | 6 | 1 | 5 | 15
  Italy | 3 | 12 | 4 | 17 | 36
  Japan | 25 | 47 | 8 | 43 | 123
  Latvia | 8 | 10 | 3 | 8 | 29
  Lithuania | 6 | 4 | 5 | 7 | 22
  Malaysia | 0 | 3 | 0 | 3 | 6
  Mexico | 1 | 3 | 2 | 4 | 10
  Netherlands | 1 | 6 | 0 | 3 | 10
  Poland | 15 | 32 | 13 | 62 | 122
  Romania | 4 | 2 | 0 | 8 | 14
  Russia | 19 | 36 | 16 | 29 | 100
  Serbia | 1 | 9 | 4 | 7 | 21
  Slovakia | 6 | 7 | 1 | 7 | 21
  South Korea | 3 | 8 | 1 | 13 | 25
  Spain | 1 | 6 | 4 | 9 | 20
  Switzerland | 0 | 4 | 0 | 6 | 10
  Taiwan | 1 | 1 | 0 | 1 | 3
  Turkey | 0 | 5 | 2 | 1 | 8
  Ukraine | 18 | 31 | 16 | 28 | 93
  United Kingdom | 2 | 4 | 2 | 6 | 14
  United States | 21 | 45 | 10 | 64 | 140

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Clinical Remission at Week 40
Description: Clinical remission at week 40 is defined as achieving a 9-point modified Mayo score for rectal bleeding=0, stool frequency=0 or 1 with ≥ 1 point decrease from baseline, and endoscopy=0 or 1 (excluding friability).
  Stool Frequency Subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); Rectal Bleeding Subscore, based on the participant's diary and scored from 0 (no blood) to 3 (blood only passed); Endoscopy Subscore, based on central reading of colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
Time Frame: Week 40
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least one dose of study drug and who had the modified Mayo score measured correctly at baseline. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 25.1 [18.8 to 31.5] | 49.9 [44.7 to 55.0]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 23.2, 95% CI 2-sided [15.2 to 31.2]

2. Secondary Outcome: Percentage of Participants in Endoscopic Remission at Week 40
Description: Endoscopic remission at week 40 is defined as achieving a Mayo endoscopic subscore of 0 or 1 (excluding friability) at Week 40. Endoscopy subscore is based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding, ulceration).
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 29.1 [22.4 to 35.7] | 58.6 [53.6 to 63.7]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.5, 95% CI 2-sided [20.2 to 36.8]

3. Secondary Outcome: Percentage of Participants With Histologic Remission at Week 40
Description: Histologic remission was assessed using the Geboes histologic scoring system developed for assessment of histologic disease activity in ulcerative colitis. Remission was defined as Geboes histological subscore of 0 for grades: 2b (lamina propria neutrophils), and 3 (neutrophils in epithelium), and 4 (crypt destruction), and 5 (erosion or ulceration).
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 24.6 [18.3 to 30.9] | 48.5 [43.4 to 53.6]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 22.5, 95% CI 2-sided [14.5 to 30.5]

4. Secondary Outcome: Percentage of Participants in Symptomatic Remission at Week 40
Description: Symptomatic remission at week 40 is defined as a Mayo score for rectal bleeding=0, stool frequency=0 or 1 with ≥ 1 point decrease from baseline.
  Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal).
  Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed).
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 39.7 [32.5 to 46.8] | 71.0 [66.3 to 75.6]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.2, 95% CI 2-sided [21.9 to 38.6]

5. Secondary Outcome: Percentage of Participants in Endoscopic Response at Week 40
Description: Endoscopic response at week 40 is defined as achieving at least a 1 point decrease from baseline in the Mayo endoscopic subscore.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 40.8 [33.6 to 48.0] | 72.6 [68.0 to 77.2]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 31.0, 95% CI 2-sided [22.4 to 39.6]

6. Secondary Outcome: Percentage of Participants in Clinical Response at Week 40
Description: Clinical response at week 40 is defined as a decrease in the 9-point modified Mayo score (MMS) [rectal bleeding, stool frequency and the endoscopic findings] inclusive of >= 2 points and >=30% from baseline with either a decrease of rectal bleeding subscore of >=1 or rectal bleeding subscore of 0 or 1.The MMS is a composite score of ulcerative colitis disease activity calculated as the sum of three subscores: Stool frequency subscore, based on the participant's diary and scored from 0 (normal number of stools) to 3 (5 or more stools than normal); Rectal bleeding subscore, based on the participant's diary and scored from 0 (no blood seen) to 3 (blood alone passed); Endoscopy subscore, based on colonoscopy or sigmoidoscopy and scored from 0 (normal or inactive disease) to 3 (severe disease, spontaneous bleeding,ulceration).
Time Frame: Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 49.2 [41.8 to 56.5] | 80.3 [76.2 to 84.4]
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 30.6, 95% CI 2-sided [22.3 to 38.9]

7. Secondary Outcome: Change From Baseline to Week 40 in Health Related Quality of Life: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score
Description: The IBDQ is a 32-item participant-completed questionnaire that measures 4 aspects of subjects' lives: symptoms directly related to the primary bowel disturbance, systemic symptoms, emotional function, and social function. Responses are graded on a 7-point. Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." Scores range from 32 to 224; a higher score indicates a better quality of life. Least square (LS) Mean was calculated using analysis of covariance (ANCOVA) model for post-baseline measures: The ANCOVA model includes: treatment, baseline value, prior biologic or tofacitinib failure (yes/no), clinical remission status (yes/no) at AMAN Week 12, and region (North America/Europe/Other).
Time Frame: Induction Baseline, Week 40
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline IBDQ measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
score on a scale | 24.51 (2.767) | 49.75 (2.102)
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with modified baseline observation carried forward (mBOCF); LS Mean difference (Final Values) = 25.24, 95% CI 2-sided [19.16 to 31.32], Standard Error of Mean 3.094

8. Secondary Outcome: Change From Baseline to Week 40 in Fecal Calprotectin
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation. Least square (LS) Mean was calculated using ANCOVA model for post-baseline measures: The ANCOVA model includes treatment, baseline value, prior biologic or tofacitinib failure (yes/no), corticosteroid use (yes/no) at AMAN baseline, region (North America/Europe/Other), Clinical Remission status (yes/no) at AMAN Week 12.
Time Frame: Induction Baseline, Week 40
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline fecal calprotectin measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: milligram per kilogram (mg/kg)
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
milligram per kilogram (mg/kg) | -1155.82 (221.394) | -1995.47 (172.443)
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with modified baseline observation carried forward (mBOCF); LS Mean difference (Final Values) = -839.64, 95% CI 2-sided [-1323.08 to -356.21], Standard Error of Mean 245.990

9. Secondary Outcome: Change From Baseline to Week 40 in Bowel Urgency Based on the Urgency Numeric Rating Scale (NRS)
Description: The Urgency NRS is a single participant reported item that measures the severity for the urgency (sudden or immediate need) to have a bowel movement in the past 24 hours using an 11-point NRS ranging from 0 (no urgency) to 10 (worst possible urgency). Higher scores indicate more severe urgency. Least square (LS) Mean was calculated using mixed model repeated measures (MMRM) model for post-baseline measures: The MMRM model includes treatment, baseline value, visit, interaction of baseline value-by-visit, interaction of treatment-by-visit, prior biologic or tofacitinib failure (yes/no), baseline corticosteroid use (yes/no), clinical remission status (yes/no) at AMAN Week 12, and region (North America/Europe/Other).
Time Frame: Induction Baseline, Week 40
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least 1 dose of study drug and had a baseline and at least one post-baseline urgency NRS measurement. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 104 | 316
score on a scale | -2.74 (0.202) | -3.80 (0.139)
Statistical Analysis 1: Comparison: Maintenance Period: Miri IR - PBO SC vs Maintenance Period: Miri IR - 200 mg Miri SC; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -1.06, 95% CI 2-sided [-1.51 to -0.61], Standard Error of Mean 0.228

10. Secondary Outcome: Percentage of Participants Hospitalized for Ulcerative Colitis (UC)
Description: Percentage of participants hospitalized for UC. Only hospitalizations associated with an adverse event with >=24 hours stay were recorded.
Time Frame: Week 40
Population: Modified Intention-to-treat population (mITT): All randomized participants who received at least one dose of study drug. Participants were analysed per their assigned treatment arm regardless of the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC
Number analyzed (Participants) | 179 | 365
percentage of participants | 1.1 | 0

11. Secondary Outcome: Pharmacokinetics (PK): Clearance of Mirikizumab
Description: Clearance of mirikizumab was evaluated.
Time Frame: Predose: Weeks 0, 4, 12, 24 and 40
Population: All randomized participants who received at least one dose of study drug subcutaneously (both induction responders and nonresponders) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour (L/h)
Groups:
- 200 Milligram (mg) Miri SC: Participants who received 200 mg mirikizumab SC every Q4W.
Arm/Group | 200 Milligram (mg) Miri SC
Number analyzed (Participants) | 652
Liters per Hour (L/h) | 0.0487 (54)

ADVERSE EVENTS:
Time Frame: Up To 40 Weeks
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Maintenance Period: Miri IR - PBO SC | Maintenance Period: Miri IR - 200 mg Miri SC | Maintenance Period: PBO IR - PBO SC | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV | Extended Induction: Induction Nonresponders - 300mg Miri IV | Open Label Maintenance: Delayed Responders - 200 mg Miri SC
All-Cause Mortality (participants affected / at risk) | 1/192 | 0/389 | 0/135 | 0/90 | 0/461 | 0/271
Serious Adverse Events (participants affected / at risk) | 15/192 | 13/389 | 7/135 | 3/90 | 21/461 | 8/271
Other Adverse Events (participants affected / at risk) | 57/192 | 90/389 | 37/135 | 13/90 | 44/461 | 54/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Maintenance Period: Miri IR - PBO SC (N=192) | Maintenance Period: Miri IR - 200 mg Miri SC (N=389) | Maintenance Period: PBO IR - PBO SC (N=135) | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV (N=90) | Extended Induction: Induction Nonresponders - 300mg Miri IV (N=461) | Open Label Maintenance: Delayed Responders - 200 mg Miri SC (N=271)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maculopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 2 (2)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacillus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurologic somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 1/160 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colectomy total (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinopexy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maintenance Period: Miri IR - PBO SC (N=192) | Maintenance Period: Miri IR - 200 mg Miri SC (N=389) | Maintenance Period: PBO IR - PBO SC (N=135) | Loss of Response (LOR) Rescue Period:LOR Cohort-300 mg Miri IV (N=90) | Extended Induction: Induction Nonresponders - 300mg Miri IV (N=461) | Open Label Maintenance: Delayed Responders - 200 mg Miri SC (N=271)
Anaemia (Blood and lymphatic system disorders) | 9 (12) | 8 (8) | 8 (11) | 5 (5) | 7 (7) | 9 (9)
Colitis ulcerative (Gastrointestinal disorders) | 35 (35) | 26 (30) | 17 (18) | 0 (0) | 4 (4) | 10 (11)
Nasopharyngitis (Infections and infestations) | 11 (11) | 28 (38) | 9 (12) | 1 (1) | 15 (15) | 14 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 26 (27) | 4 (4) | 3 (5) | 15 (15) | 19 (24)
Headache (Nervous system disorders) | 2 (5) | 16 (21) | 5 (18) | 5 (5) | 8 (10) | 13 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/92/NCT03524092/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03524092/SAP_001.pdf